CLINICAL TRIAL: NCT05179811
Title: Description of the Evolution of Functional Dysphonia Managed by Hypnotherapy
Acronym: HYPNODYS
Status: Terminated | Type: Observational
Why Stopped: lack of recrutement
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: CHH_2021_22
Record Dates: First submitted 2021-09-10; First posted 2022-01-05 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Functional Dystonia (Disorder)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Patients with functional dysphonia using the Voice Handicap Index score.
  Interventions: Procedure: Hypnosis sessions

INTERVENTIONS:
Procedure: Hypnosis sessions — * Physical examination
  * Psychiatric Assessment
  * VHI, SF-36, IPQ-R questionnaires
  * Standardized voice recording
  * 3 Standardized Hypnotherapy sessions
  * CGI-I-Patient Questionnaire

SUMMARY:
HYPNODYS is a single-center study evaluating the evolution of perceived voice-related disability before and after 3 standardized hypnosis sessions in patients with functional dysphonia.

DETAILED DESCRIPTION:
Functional or psychogenic voice and speech disorders are characterized by various changes in voice (aphonia or dysphonia) or speech (stuttering, foreign accent syndrome, and childish prosody in adults) without organic damage associated. These disorders have a significant functional impact (physical and mental handicap) and a significant cost for society.

Their management, like that of functional neurological disorders in general, is still poorly codified. Different therapeutic strategies are mentioned, especially in the event of speech therapy failure, in particular behavioural and cognitive psychotherapeutic approaches.

The recent explanatory hypotheses of functional neurological disorders are that the processing of sensory and motor information can be modulated, or even inhibited, by cognitive and attentional mechanisms. Different elements (volition, emotions, attention) can exclude certain psychic representations from consciousness.

Hypnosis, by exercising direct control over attentional resources makes it possible to obtain hypoactivation of the medial prefrontal cortex and hyperactivation of the executive and salience networks, making greater use of the buffer of working memory and activate the para-sympathetic system. Thus, one can observe analgesia, amnesia, a loss of the notion of time, plurimodal hallucinations, a detachment from oneself, a distortion of reality and logic.

Hypnosis has been used since the 19th century in the treatment of functional paralysis. To date, there are only presentations and case series evaluating the value of hypnosis in functional disorders of voice and speech. However, from a clinical standpoint, the use of hypnosis seems to show a significant interest in functional speech disorders.

Functional neurological disorders are located at the crossroads of neurological and psychiatric disorders, psychiatric and psychological evaluation of these patients therefore seems necessary in order to measure their impact on the pathological and recovery processes through hypnotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of functional neurological disorder according to the DSM-5
* Supported at the Rothschild Foundation as part of a hypnotherapy protocol
* Mastering the understanding of the French language
* Express consent to participate in the study

Exclusion Criteria:

* Organic etiology of dysphonia
* Decompensation of a psychiatric pathology
* Discovery during study of an organic etiology not initially identified

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with functional dysphonia using the Voice Handicap Index score
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Evolution of perceived voice related disability before and after 3 standardized hypnosis sessions | day 0 and 3 months after last hypnosis session
  Description of this evolution using the Voice Handicap Index score VHI.The questionnaire items were grouped into three equal parts which represent three aspects of voice disorders: functional, emotional and physical. The Voice Handicap Index consists of 30 items, or 10 items per game. The questionnaire is completed item by item by choosing one of the following five answers according to frequency: never, almost never, sometimes, almost always and always.The scores assigned to the answers range from zero to four points, knowing that never is zero and always is worth. The average of the total score at VHI obtained by so called normal subjects, without voice disturbance, is 6.86. A subject obtaining a score equal or less than 6.86 does not present a vocal handicap. A score greater than or equal to 26.62 is pathological

CONTACTS AND LOCATIONS:
Overall Officials: Cécile HUBSCH, Principal Investigator — Hôpital Fondation A. de Rothschild; Stéphane MOUCHABAC, Study Director — Hôpital Saint-Antoine
Locations (1):
- Hôpital Fondation A. de Rothschild, Paris, France